CLINICAL TRIAL: NCT04161677
Title: Mitigation Investigation for Spinal Manipulation Treatments (MIST) - Part 3: Continued Assessment & Feasibility of an Electronic Active Surveillance Reporting System
Brief Title: MIST3: Active Patient Safety Reporting
Acronym: MIST3
Status: Completed | Type: Observational
Sponsor: Parker University (Other)
Responsible Party: Sponsor
Other Study IDs: Parker19_05
Record Dates: First submitted 2019-11-10; First posted 2019-11-13 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Safety Issues
Keywords: Adverse event; Electronic reporting system; Chiropractic; Spinal manipulation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will seek to describe and understand adverse events (AE) severity ratings.

DETAILED DESCRIPTION:
Using an explanatory mixed methods design, three different quantitative methods 1. severity ratings based on a series of questions, 2. severity rating based on severity terms, and 3. severity based on definitions will be used to conduct a feasibility study on understanding adverse event reporting system.

ELIGIBILITY:
Inclusion Criteria:

* Health patients

Exclusion Criteria:

* None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A convenience sample of all patients at the Parker University Wellness clinic will be invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Pre-screening questionnaire | 5-10 minute
  Severity rating based on a series of questionnaire
Post-survey | Immediately after visit
  Severity rating based on severity term questionnaire
follow-up questionnaire | 7-10 days after visit
  Severity rating based on definitions questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Parker University, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided